CLINICAL TRIAL: NCT05495256
Title: Monitoring Metered Dose Inhalation (MDI) Volume and Timing With a Respimetrix Device in Obstructive Lung Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonary Critical Care Associates of Baltimore (Other)
Collaborators: Gerresheimer (Unknown)
Responsible Party: Principal Investigator, Alan Schwartz, Principal Investigator, Pulmonary Critical Care Associates of Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Respimetrix 2
Record Dates: First submitted 2022-04-19; First posted 2022-08-10 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Asthma; Copd
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: patients are screened, consented, and all go through the inhaler training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- MDI Training (Other): All participants are led through the MDI training with the Respimetrix Device. Protocol is within groups design.
  Interventions: Device: Respimetrix

INTERVENTIONS:
Device: Respimetrix — The Respimetrix device has a low resistance airflow sensor with an inhaler to measure patients inspiratory airflow and volume. This device will thereby provide quantifiable measures of lung function and bronchodilator delivery.

SUMMARY:
To Determine whether use of the Respimetrix flow test device a) can determine "good" versus "poor" inhaler techniques, and b) the effects of the inhaler training on technique.

DETAILED DESCRIPTION:
Good metered dose inhaler (MDI) technique is described as sitting or standing upright with the head slightly tilted back, exhaling fully, and then inhaling slowly and deeply as you activate the MDI. Common mistakes include: not exhaling fully; not inhaling deeply enough; inhaling too quickly, and not activating the MDI at the proper time.

This study will use the Respimetrix device with placebo to assess a patient's inhaler technique, provide training to patients who demonstrate poor inhaler technique, and remotely track a subject's breathing ability over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Current diagnosis of asthma or Chronic obstructive pulmonary disease (COPD) patients
* Patients must be willing and able to provide informed consent to participate in the the study.
* Patients must be able to use a metered dose inhaler

Exclusion Criteria:

* Contraindication to inhaler use
* Tracheostomy
* Incapacitating disability that interferes with the use of the inhaler or execution of the protocol
* Unable to understand informed consent (e.g. non-English speakers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Change in pressurized metered-dose inhaler (pMDI) performed after training using Respimetrix device | 2 weeks
  Measure actuation timing, flow rate and volume after intervention

SECONDARY OUTCOMES:
Describing baseline pressurized metered-dose inhaler (pMDI) technique | 2 weeks
  Measure actuation timing, flow rate and volume before intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Pulmonary and Critical Care Associates Of Baltimor, Towson, Maryland, United States

IPD SHARING:
Plan to Share IPD: No